CLINICAL TRIAL: NCT05662514
Title: Effect of Probiotics on Gut Microbiota During the Helicobacter Pylori Eradication: a Randomized Double-blind Placebo-controlled Trial
Brief Title: Effect of Probiotics on Gut Microbiota During the Helicobacter Pylori Eradication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KYLL-202210-011
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-12

CONDITIONS: Helicobacter Pylori Infection; Gut Microbiota
Keywords: Helicobacter pylori; Gut microbiota; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Esomeprazole 20 mg and bismuth 2g twice daily before meals, amoxicillin 1 g, and clarithromycin 500 mg twice daily after meals, probiotic once a day with one packet each time 2 hours after taking medicine above in the evening, for 2 weeks.
  Interventions: Dietary Supplement: Bifidobacterium animalis subsp. lactis BLa80
- Placebo group (Placebo Comparator): Esomeprazole 20 mg and bismuth 2g twice daily before meals, amoxicillin 1 g, and clarithromycin 500 mg twice daily after meals, placebo once a day with one packet each time 2 hours after taking medicine above in the evening, for 2 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium animalis subsp. lactis BLa80 — Test product contain 3 × 109 colony-forming units [CFU] Bifidobacterium animalis subsp. lactis BLa80 strains, for each packet.
  Subjects ingested one packet (3 g/packet) of Test product per day (2 hours after taking antibiotics in the evening), for 14 days.
  Arms: Probiotic group
Other: Placebo — To maintain the blinding, patients in the control group received placebo included in identical packets. Control product per day (2 hours after taking antibiotics), for 14 days.
  Arms: Placebo group

SUMMARY:
Helicobacter pylori (H. pylori) is still infecting more than half of the population in many countries, although the prevalence is decreasing. As a main cause of chronic gastritis, peptic ulcer, and malignant gastric tumors, H. pylori places a heavy burden on developing countries and regions with high infection rate. In the last decade, the eradication rates of conventional regimens based on proton pump inhibitors (PPIs) plus antibiotics have been decreasing. Antibiotic resistance and decrease of drug compliance caused by adverse effects were the two main reasons for eradication failure. Moreover, H. pylori treatment causes dysbiosis of gut microbiota and increases the expression of antibiotic resistance gene. Therefore, eradication of H. pylori is facing a great challenge, and effective and safe methods are needed.

To reduce adverse effects, improve drug compliance and increase eradication rates, certain probiotics were added to conventional regimens in several clinical studies. Probiotics were more or less shown to reduce adverse effects in the vast majority of clinical studies, but whether probiotics can improve the eradication rate of H. pylori remains controversial. Meanwhile, several studies focusing on the impact of probiotics on gut microbiota during H. pylori eradication have been published recently. Thus, we conducted a randomized, double-blind, placebo-controlled trial aiming to evaluate the effects of probiotics combining with 14-day bismuth quadruple therapy on H. pylori eradication.

DETAILED DESCRIPTION:
This was a randomized, parallel-group, double-blind and placebo-controlled study. If the subject meets the selection criteria but not the exclusion criteria, and signs an informed consent form, patients were randomly allocated in a 1:1 ratio to receive either the investigational product or placebo along with H. pylori eradication therapy. The randomization sequence was generated using SAS 9.1.3. Eight weeks after the eradication treatment, the subjects will review the 13C-urea breath test, and the researcher records the results. Feces samples, which were taken at the subject's home at the beginning, the end of treatment and 8 weeks after treatment completion, were collected from the patients immediately and stored at -80 °C until analysis. In this study, the influences of antibiotics and combination of probiotics on gut microbiota during H. pylori treatments were investigated using high-throughput sequencing of the 16S rRNA gene.

Patients were required to recall the history of gastrointestinal symptoms at baseline, keep the symptom diaries during the treatment and return the diaries at week 2. Gastrointestinal symptoms were assessed and scored according to the 15-iteem GSRS27 before (week 0) and after quadruple therapy (week 2). Special attention was given to the following symptoms: epigastric pain, heartburn, acid regurgatition, nausea or/and vomiting, abdominal distension, eructation, diarrhea, constipation. Adverse effects outside gastrointestine were also recorded and evaluated.

Compliance with antibiotic therapy and the investigational product was evaluated by means of a patient's diary and product accountability, while compliance with eradication therapy was evaluated through a questionnaire. After all subjects were tested, the eradication rates, adverse reaction rates and patient compliance of each group were calculated.

Patients were evaluated at 4 visits: screening (10-30 days before the baseline visit), baseline, end of treatment/efficacy (14 days after the baseline visit) and follow-up (8 weeks after treatment completion). Patients were diagnosed with one (or more) of three validated methods, 13C-urea breath test, rapid urease test or histology, depending on the clinical situation of the patient. Eradication confirmation test was also performed following standard recommendations: 13C-urea breath test at 8 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-70.
2. Patients with H. pylori infection (Positive for rapid urease test or 13C/14C-urea breath test).
3. Patients who have did not receive H. pylori eradication treatment before.

Exclusion Criteria:

1. Patients with serious underlying diseases, such as liver insufficiency (Aspartate aminotransferase or alanine aminotransferase greater than 1.5 times the normal value), renal insufficiency (Cr≥2.0mg/dL or glomerular filtration rate <50 ml/min), immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.
2. Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.
3. Patients with active gastrointestinal bleeding.
4. Patients with a history of upper gastrointestinal surgery.
5. Patients allergic to treatment drugs.
6. Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs which might influence gut microbiota within 3 months.
7. Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse.
8. Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota | Week 0, week 2 and week 10
  Stool samples were collected at wk0, wk2, and wk10. Patients were instructed to collect stool samples at the medical visit site by using disposable sterile feces collection tubes. Samples were stored at -80℃ after collection immediately. In this study, the influences of antibiotics and combination of probiotics on gut microbiota during H. pylori treatments were investigated using high-throughput sequencing of the 16S rRNA gene.

SECONDARY OUTCOMES:
Rate of adverse reactions | Week 2 and week 10
  Rate of adverse reactions
Patient compliance | Week 10
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhou, Dr, Study Chair — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang C, Liang L, Lv P, Liu L, Wang S, Wang Z, Chen Y. Effects of non-viable Lactobacillus reuteri combining with 14-day standard triple therapy on Helicobacter pylori eradication: A randomized double-blind placebo-controlled trial. Helicobacter. 2021 Dec;26(6):e12856. doi: 10.1111/hel.12856. Epub 2021 Oct 10. PMID 34628695
- [Background] Yuan Z, Xiao S, Li S, Suo B, Wang Y, Meng L, Liu Z, Yin Z, Xue Y, Zhou L. The impact of Helicobacter pylori infection, eradication therapy, and probiotics intervention on gastric microbiota in young adults. Helicobacter. 2021 Dec;26(6):e12848. doi: 10.1111/hel.12848. Epub 2021 Aug 26. PMID 34448282
- [Background] Nabavi-Rad A, Sadeghi A, Asadzadeh Aghdaei H, Yadegar A, Smith SM, Zali MR. The double-edged sword of probiotic supplementation on gut microbiota structure in Helicobacter pylori management. Gut Microbes. 2022 Jan-Dec;14(1):2108655. doi: 10.1080/19490976.2022.2108655. PMID 35951774
- [Result] Guillemard E, Poirel M, Schafer F, Quinquis L, Rossoni C, Keicher C, Wagner F, Szajewska H, Barbut F, Derrien M, Malfertheiner P. A Randomised, Controlled Trial: Effect of a Multi-Strain Fermented Milk on the Gut Microbiota Recovery after Helicobacter pylori Therapy. Nutrients. 2021 Sep 11;13(9):3171. doi: 10.3390/nu13093171. PMID 34579049